CLINICAL TRIAL: NCT06919783
Title: Adapting a Health at Every Size Intervention to Obstetric Care
Acronym: OB-HAES
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Anna Whelan, Assistant Professor in Obstetrics and Gynecology, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0001474; 5KL2TR1455-8 (Other Grant/Funding Number: UMass Chan Center for Clinical and Translational Science); 5KL2TR001455 (NIH)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Weight Stigma
Keywords: weight stigma; health at every size; perinatal mood disorders; perinatal anxiety; perinatal depression; postpartum anxiety; postpartum depression; eating disorders; pregnancy
MeSH Terms: conditions — Weight Prejudice; Depression, Postpartum; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OBHAES Intervention (Experimental): Individuals will be invited to participate in 5 group sessions in pregnancy and the postpartum period. The sessions include education on pregnancy, mental health, nutrition, and self-advocacy.
  Interventions: Behavioral: Health at Every Size in Obstetrics

INTERVENTIONS:
Behavioral: Health at Every Size in Obstetrics — Individuals are invited to participate in 5 group sessions during pregnancy and the postpartum period. The sessions will last 2-2.5 hours each and will include education on pregnancy, mental health, nutrition, movement, and self-advocacy. The sessions will be administered by an OBGYN/MFM physician and psychologist and include discussion with doulas, registered dieticians with pregnancy and disordered eating experience, and prenatal yoga instructors.

SUMMARY:
Perinatal mental health disorders occur in 1 in 5 pregnancies and have significant negative intergenerational consequences including being the leading cause of overall and preventable mortality during pregnancy and the first year postpartum. Perinatal mental health disorders impact not only the individual but can also have adverse effects on immediate and long-term child and family wellbeing. Untreated mental health disorders in pregnancy are associated with preterm birth, low birth weight, impaired bonding and lead to issues with neonatal neurodevelopment. Interventions to prevent perinatal mental health disorders are of the utmost importance in helping to improve maternal and child health outcomes in the United States.

In Massachusetts, almost a quarter of pregnant people have a BMI >30 kg/m2. Rates of perinatal mental health disorders are higher among individuals with elevated body mass index (BMI) > 30 kg/m2 compared to people with BMI < 30 kg/m2. People with BMI > 30 are 50% more likely to have antenatal depression, 40% more likely to have postpartum depression, and 25% more likely to develop postpartum anxiety compared to those with BMI <30 kg/m2. The etiology for the increased risk for perinatal mental health disorders among persons with a higher BMI has not been extensively investigated. However, some postulate this could be due to an increase in the medicalization of pregnancy, along with complications for the birthing person or with fetal/neonatal health. Over the last few years, some researchers have begun to hypothesize that weight stigma may also play a significant role in the development of perinatal mental health disorders in this population.

Weight stigma - the social rejection and devaluing of people who live in bodies which do not conform to the societal standards of weight - is associated with the development of depression among people with BMI >30. Weight stigma has been demonstrated through many fields of healthcare. Many providers hold beliefs regarding people with elevated BMIs, including that they are lazy and unintelligent. Providers may also blame individuals for their medical complications and are less likely to offer them interventions including surgery. This leads to worse outcomes and people avoiding care. Additionally, external weight stigma can lead to weight bias internalization, where individuals accept and self-direct negative stereotypes toward themselves.

Weight stigma leads to a cycle of internalized bias which is then compounded by traumatic experiences of stigmatization by healthcare providers. This may lead patients to avoid care and be at increased risk for adverse health outcomes (include adverse mental health outcomes). In fact, the American Association of Endocrinology recommends incorporating the experience of bias and stigmatization into the diagnosis and staging of obesity. Therefore, one could postulate that weight stigma and weight bias internalization likely contribute to the high prevalence of perinatal mental health conditions among individuals with elevated BMI.

In order to combat weight stigma and weight bias internalization in people seeking healthcare, the Association for Size Diversity and Health created the Health at Every Size (HAES) intervention. HAES characterizes health as a continuum that is specific to the individual and varies with time and circumstance. HAES has five principles including weight inclusivity, health enhancement, eating for well-being, respectful care, and life enhancing movement. Previously studied HAES interventions consist of a number of group sessions led by trained clinicians that are based on these principles. The sessions range in topics from nutrition, physical activity, self-efficacy and acceptance in order to decrease internalization of weight bias.

Previous data from the primary care literature demonstrates the efficacy of HAES interventions on improving overall well-being, decreasing rates of depression and other mental health disorder symptoms, and even in improving cardiovascular and lipid profiles.

Despite these findings, HAES has not yet been adapted for use in an obstetric context despite the traditional model for prenatal care being highly focused on weight. Patients are weighed at each prenatal visit, and the amount of "appropriate" weight gain is calculated based on BMI. People with an elevated BMI receive extra laboratory testing, ultrasounds and fetal monitoring. This almost extreme perseverance on weight during pregnancy causes individuals in larger bodies to experience significant weight stigma during their prenatal care.

Obstetric providers and perinatal people are interested in interventions to assist in the provision of sensitive care for people who experience weight stigma. This project aims to utilize patient and expert input to adapt a HAES intervention to an obstetric context (OB-HAES).

DETAILED DESCRIPTION:
After written informed consent is obtained, participants will be enrolled in the OB-HAES intervention (N=10). They will complete demographic questionnaires as well as weight bias internalization scale (WBIS) , prenatal eating disorder behavior scale and everyday discrimination scale (EDDS). Participants will come to in-person group sessions in addition to their routine obstetric care. These sessions will be held in the evening (after working hours). Similar to the set-up of Centering Pregnancy, in addition to the group support and educational activities, an obstetric and psychiatry provider will be available following the meeting to discuss and urgent concerns that participants have and to assist in coordination if further care is required. After each session, participants will complete surveys on REDCap regarding acceptability and feasibility of the session. After the 5th and final session which occurs in the post-partum period, participants will be scheduled for interviews regarding their experience and feedback of the program. They will also be sent a REDCap survey link to complete WBIS, EDD and assessment of perinatal mood and anxiety disorders (EPDS and GAD-7). Information regarding participants medical history, pregnancy and delivery outcomes will be abstracted from the medical records. Based on the feedback from Phase 1, we will offer participants the option to have partner accompany them during group sessions in Phase 2. We will provide fact sheets to the partners and obtain their verbal consent.

Phase 2 will consist of five two-hour group sessions conducted by Drs Whelan and Williams from the research team with assistance from multidisciplinary experts as follows:

Session 1 will be focused on introductions to pregnancy/prenatal care timeline, importance of mental health care, and introduction to Health at Every Size. Dr. Williams will begin the session discussing mental health and the connection of mental health to physical health and lead participants through a mindfulness/grounding exercise. Drs Whelan and Williams will then discuss Health at Every Size as guiding principles for healthcare and how they can be used to improve participants relationship with food, activity and their bodies. There will be a snack and bathroom break followed by information on what to expect over the course of pregnancy/prenatal care and question and answer session led by Dr. Whelan. Since we are aiming to improve the overall health of participants, we plan to distribute handouts on how to self-monitor blood pressure (BP) at home and provide them with a portable BP apparatus during the session. Additional handouts will also be distributed during each session.

Session 2 will be centered on nutrition and movement during pregnancy. After Dr. Williams leads the group in a mindfulness exercise, Sarah Anzlovar RD will share information about nutrition during pregnancy. Sarah Anzlovar is a registered dietician with expertise working with perinatal individuals and uses a Health at Every Size framework for her care. She has helped develop educational information and will be leading part of session 2 but will not be engaging in research activity. The nutrition portion of the class will be followed by a snack and break during which Dr. Whelan will speak about screening for and treating gestational diabetes.

The second half of session 2 will be a prenatal yoga/stretching activity lead by Hari Kirin Khalsa and Jayna Turchek. Khalsa and Turchek are yoga instructors who specialize in developing perinatal adaptive yoga for mind-body connection. They will lead two sessions throughout the intervention but will not be engaging in research activities.

Participants are expected to sign a waiver to participate in the yoga session.

The third session is focused on external and internalized weight bias and self-advocacy. Dr Williams will help the group focus by leading them through a grounding exercise. Dr. Whelan and Dr. Williams will then facilitate a group discussion of participant experience of living in a larger body and navigating pregnancy/the healthcare system. Dr. Williams will then lead the group through a dialectical behavioral activity which helps individuals learn tools for boundary setting. After this activity there will be a break/snack. After the break participants will hear from two doulas about how a doula can support and advocate for them during pregnancy and labor. Cheyenne Bell and Amber Matteson are doulas with multiple years of experience supporting pregnant people, particularly those marginalized due to their race/ethnicity and body size. They will lead this portion of the intervention but will not be engaging in research activities.

The fourth session is the final session prior to the participants giving birth. This session will again open with mindfulness by Dr. Williams and then the majority of the time will be educational information about labor and delivery, mode of delivery, and the monitors/instruments used to assist in care led by Dr. Whelan. Participants will have the opportunity to touch and see external and internal monitors. After break, the participants will be joined again by Cheyenne Bell and Amber Matteson to help discuss pain control and options for non-pharmacologic labor management. The participants will then spend time developing a birth plan with the assistance of Dr. Whelan, Cheyenne Bell and Amber Matteson. Cheyenne Bell and Amber Matteson will not be engaging in any research activities.

The final session will occur in the postpartum period. Participants and their newborns will be invited back. Dr. Williams will facilitate a mindfulness activity and then Dr. Whelan and Williams will facilitate a group discussion of all individuals birth and postpartum experiences. They will also share information on community resources for new parents. Hari Kirin Khalsa and Jayna Turchek will also return to discuss movement in the postpartum period and lead the participants through some stretching activities.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are between 18 and 50 years of age, have a BMI >30 kg/m2, and are in the first trimester of their first pregnancy.
* English speaking

Exclusion Criteria:

* Individuals who are not pregnant or do not meet inclusion criteria

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability Questionnaire | Within 2 weeks of completion of each group session.
  Eleven item questionnaire adapted from Sekhon et al (BMC Health Service Research 2022). This questionnaire will ask participants to rate the acceptability of the intervention including how comfortable they were participating, how what they learned may help them, as well as identify areas for improvement in the intervention and roadblocks.

SECONDARY OUTCOMES:
Qualitative Interviews | within 6 weeks of final session
  Participants will be asked to complete qualitative interviews about their experience with the OB-HAES intervention following the completion of the final group session.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Whelan, MD, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This data would be identifiable as there are so few planned participants.